CLINICAL TRIAL: NCT01050426
Title: A Multicentre Randomised Phase II Clinical Study of UFT/Leucovorin, Radiotherapy With or Without Cetuximab Following Induction Gemcitabine Plus Capecitabine in Patients With Locally Advanced Pancreatic Cancer (PERU)
Brief Title: A Clinical Study of UFT/Leucovorin, Radiotherapy With or Without Cetuximab Following Induction Gemcitabine Plus Capecitabine in Patients With Locally Advanced Pancreatic Cancer (PERU)
Acronym: PERU
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data from other trials failed to demonstrate meaningful survival advantage
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3065
Record Dates: First submitted 2009-12-21; First posted 2010-01-15 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Tegafur; Leucovorin; Cetuximab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): UFT/LV + RT
  Interventions: Other: UFT, Leucovorin
- Group 2 (Active Comparator): UFT/LV + RT + Cetuximab
  Interventions: Other: UFT/ Leucovorin + Cetuximab + Radiotherapy

INTERVENTIONS:
Other: UFT, Leucovorin — UFT 300mg/m2/day in 3 equal doses and Leucovorin 90mg/day in 3 divided doses per day given daily on the days of radiotherapy only (30 days in total)
  Arms: Group 1
Other: UFT/ Leucovorin + Cetuximab + Radiotherapy — UFT 300mg/m2 + LV 90mg/day on days of RT only (30 days in total), Cetuximab 400mg/m2 week 1, thereafter 250mg/m2 weeks 2-6
  Arms: Group 2

SUMMARY:
The purpose is to assess the overall survival of patients receiving either UFT/LV + radiotherapy (RT) or UFT/LV + Cetuximab + RT after neo-adjuvant chemotherapy.

DETAILED DESCRIPTION:
Locally advanced pancreatic cancer carries a poor prognosis with no survival advantage of CRT over chemotherapy alone. 4 Phase II- III studies patients without disease progression after 3 months of systemic chemotherapy and CRT had a longer survival than those continuing on chemotherapy. Therefore chemotherapy followed by CRT may be a better approach. Also the effect of blocking EGFR will be evaluated in locally advanced pancreatic cancer. Gemcitabine and capecitabine combination will be used as neo-adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Histological or cytological diagnosis of adeno- or undifferentiated non-small cell carcinoma of pancreas.
* Considered to be unresectable based on following: extensive peri-pancreatic lymph node involvement, encasement or occlusion of the SMV or SMV/portal vein confluence, direct involvement of SMA, coeliac axis, inferior vena cava or aorta.
* Performance status 0-2
* No evidence of metastatic disease as determined by CT scan/ other investigations
* Adequate bone marrow function with platelets>100^9/l; WBC>3x10^9/l;neutrophils> 1.5x10^9/l
* Serum bilirubin ,1.5 x ULN and transaminases < 2.5 x ULN
* Calculated/measured GFR >50ml/min
* No concurrent uncontrolled medical condition
* No active malignant disease other than non-melanotic skin cancer or carcinoma in situ of the uterine cervix over the last 10 years
* Life expectancy > 3months
* Adequate contraceptive precautions
* Informed written consent

Exclusion Criteria:

* medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Presence of met. disease
* Concurrent uncontrolled medical conditions
* Any previous chemo/RT or any investigational treatment for advanced pancreatic cancer.
* Adjuvant chemo + fluoropyrimidine or gemcitabine within 12months of trial entry
* Adjuvant RT with/without chemo for pancreatic cancer.
* Pregnancy/breast feeding
* Patients with known malabsorption syndromes ro a lack of physical treatment of the upper GI tract.
* Patients with a known hypersensitivity to 5-FU or with a DPD deficiency.
* Clinically significant CVD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
One year overall survival, measured from the date of registration. | one year

SECONDARY OUTCOMES:
Progression free survival | three years
Characterise safety profile of UFT/leucovorin, radiotherapy with or without cetuximab following induction gemcitabine plus capecitabine in patients with locally advanced pancreatic cancer | three years
Objective response rate | three years
Pattern of failure | up to 3 years
Quality of life | up to 3 years
Evaluation of molecular and genetic predictors of response to anti-EGFR treatment | up to 3 years
Evaluation of changes in diffusion weighted MRI parameters in pancreatic cancer patients before and after treatment. | up to 3 years
Evaluation of the role of FDG-PET in predicting overall survival, progression free survival and objective response rate in locally advanced pancreatic cancer. | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian Chau, Principal Investigator — The Royal Marsden NHS Trust
Locations (8):
- United Kingdom (8):
  - Kent Oncology Centre, Royal Tunbridge Wells, Maidstone
  - Royal Surrey County Hospital NHS Trust, Guildford, Surrey
  - The Royal Marsden NHS Trust, Sutton, Surrey
  - Aberdeen Royal Infirmary, Aberdeen
  - The Royal Bournemouth Hospital, Bournemouth
  - Christie Hospital NHS Foundation Trust, Manchester
  - Clatterbridge Centre for Oncology NHS Foundation Trust, Metropolitan Borough of Wirral
  - Poole Hospital NHS Trust, Poole